CLINICAL TRIAL: NCT02303782
Title: A Phase Ib/II Study Assessing the BET-bromodomain (BRD) Inhibitor OTX015 in Combination With Azacitidine (AZA) or AZA Single Agent in Patients With Newly-diagnosed Acute Myeloid Leukemia (AML) Not Candidate for Standard Intensive Induction Therapy (SIIT)
Brief Title: A Study Assessing tOTX015 in Combination With Azacitidine (AZA) or AZA Single Agent in Patients With Newly-diagnosed Acute Myeloid Leukemia (AML) Not Candidate for Standard Intensive Induction Therapy (SIIT)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncoethix GmbH, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8628-004; OTX015_206 (Other: OncoEthix)
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — OTX015; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OTX015 + azacitidine (Experimental)
  Interventions: Drug: OTX015; Drug: Vidaza (azacitidine)
- Azacitidine (Experimental)
  Interventions: Drug: Vidaza (azacitidine)

INTERVENTIONS:
Drug: OTX015
  Arms: OTX015 + azacitidine
Drug: Vidaza (azacitidine)

SUMMARY:
This study is designed in its first part (phase Ib) to determine the recommended dose of the OTX015 + Vidaza (azacitidine) combination in newly diagnosed acute myeloid leukemia patients not candidate for standard intensive induction therapy.

It will be followed by a randomized phase II part to assess the efficacy of the combination using 2 arms : Vidaza (azacitidine) alone vs. OTX015 in combination with Vidaza (azacitidine).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to beginning protocol-specific procedures. Patients registered for this trial must be treated and followed at the participating centers.
2. Newly-diagnosed confirmed AML, defined as > 20% myeloid blasts in the bone marrow.
3. Patients not candidate for standard intensive induction therapy (SIIT) with anthracycline and cytarabine (3+7) due to age, and/or poor general condition, and/or comorbidities, and/or any condition predicting a poor benefit/risk ratio of such chemotherapy, including complex karyotypes or secondary AML (including those with myelodysplastic features and 20-30% bone marrow blasts, who are already standard indication for AZA single agent therapy). There is no upper age limit and no protocol definition of co-morbidities. The decision that the patient is not candidate for SIIT will be made by the investigator team according to routine daily practice, based on the combination of these parameters and patient preference. The reasons for non-eligibility for SIIT will be documented in the inclusion procedures to characterize the treated population.
4. Patients > 18 years old.
5. Life expectancy of at least 3 months.
6. ECOG performance status (PS) of 0 to 2. Patients with PS > 2 at the time of diagnosis may still be enrolled, provided their PS improves to ≤2 after hematologic supportive care (transfusions, antibiotics, hydration, correction of metabolic disturbances, correction of hyperleukocytosis with hydroxyurea).
7. Patients should not have previously received other anti-leukemia drugs, except hydroxyurea (± mercaptopurine [6MP] or thioguanine [6TG]), given to control rapidly increasing hyperleukocytosis. Hydroxyurea (±6MP or 6TG) must be stopped at least 48 hours prior to start study treatment. It may be resumed to control hyperleukocytosis from Day 3 to 57. Patients who still need hydroxyurea (± 6MP or 6TG) beyond Day 57 (or end of cycle 2 in case of treatment delay) should be considered as having treatment failure.
8. Calculated creatinine clearance (CrCl) < 30 mL/min (Cockroft & Gault formula, or MDRD formula for patients aged > 65 years). Patients with CrCl < 60 mL/min should be considered at risk for increased hematologic toxicity and renal toxicity.
9. Adequate LFTs: Total bilirubin ≤ the institutional upper limit of normal (ULN); ALAT/ASAT > 3 x ULN (or > 5 x ULN in case of leukemic liver involvement).
10. Serum albumin > 28 g/L.
11. Complete baseline disease assessment workup (including routine cytogenetics and centralized assessment of molecular biomarkers) prior to the first study treatment administration.

Exclusion Criteria:

1. Pregnant or lactating women or women of childbearing potential not using adequate contraception. Male patients not using adequate contraception.
2. Patients with acute promyelocytic leukemia, or uncontrolled symptomatic disseminated intravascular coagulation (DIC).
3. Increasing or stable hyperleukocytosis > 15 G/L despite optimal hydroxyurea dose (± 6MP or 6TG).
4. Uncontrolled disease-related metabolic disorder.
5. Patients unable to swallow oral medication or with a gastrointestinal condition (e.g. malabsorption, resection) deemed to jeopardize intestinal absorption of OTX015.
6. Other serious illness or medical condition, which in the investigator's opinion could hamper understanding of the study by the patient, patient's compliance to study treatment, patient's safety or interpretation of study results. These conditions include (but are not restricted to):

   * Congestive heart failure or angina pectoris except if medically controlled, previous history of myocardial infarction within 1 year of study entry, uncontrolled hypertension or arrhythmias.
   * Significant neurologic or psychiatric disorders impairing ability to obtain consent.
   * Second cancer, needing systemic therapy.
   * Known HIV positivity, hepatitis B positivity by surface antigen expression, or active hepatitis C infection (PCR positive or antiviral therapy for hepatitis C within last 6 months).
7. Concomitant therapy with strong CYP3A4 interfering drugs.
8. Concurrent treatment with other experimental therapies or participation in another clinical trial within 21 days prior to first study treatment administration or 5 half-lives of previously administered drugs, whichever is longer, or previous anti-leukemic therapy other than hydroxyurea (± 6MP or 6TG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity occurrence for determination of Maximum Tolerated Dose | First 28 days
Complete Remission rate | at day 29
Complete Remission rate | at day 57
Complete Remission Rate | at day 115